CLINICAL TRIAL: NCT03526640
Title: Computed Tomography (CT) Guided Lung Biopsy With Plug - Evaluation of Safety and Efficacy
Brief Title: Computed Tomography (CT) Guided Lung Biopsy With Plug
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Haseem Ashraf, Associate professor, PhD, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AHUS plug study 001
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Computed Tomography, Biopsy, Pneumothorax, Chest Tube, Plug
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Intervention Model Description: Block randomized design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plug Arm (Experimental): Participants randomized for plug arm will be treated with a plug after CT guided is conducted.
  Interventions: Device: The BioSentry Tract Sealant System
- Non Plug arm (No Intervention): No Intervention, i.a. CT guided biopsy without plug.

INTERVENTIONS:
Device: The BioSentry Tract Sealant System — The BioSentry Tract Sealant System consists of a delivery system and a coaxial adapter with Bio-Seal™ plug. The hydrogel plug is deployed in the tract created by the lung biopsy needle and self-expands upon contact with moist tissue.
  Arms: Plug Arm

SUMMARY:
Protocol Title:

Computed Tomography (CT) Guided Lung Biopsy with BioSentry Plug, Evaluation of Safety and Efficacy.

DETAILED DESCRIPTION:
Protocol Summary:

Prospective, randomized, controlled, unblinded, post-market, single-center clinical study

Objectives:

Patients treated with the BioSentry system will be compared to patients not treated with the BioSentry System (Control Group).

Primary Objective:

Evaluate the rate of chest tube placement after percutaneous transthoracic needle lung biopsy

Secondary Objectives:

Evaluate the rate of intra-procedural pneumothorax Evaluate the rate of post-procedural pneumothorax Evaluate cost associated with complications Evaluate the number of hospital admissions

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to any study related procedure
2. Male or female, aged ≥18 years or older
3. Percutaneous transthoracic needle lung biopsy indicated

Exclusion Criteria:

There are no specific exclusion criteria for the study. All participants are evaluated by a pulmonologist prior to admission and determined eligible for the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2018-05-04 (Actual); Primary Completion 2020-08-04 (Estimated); Study Completion 2023-08-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the rate of chest tube | 2 years
  Evaluate the rate of chest tube placement after percutaneous transthoracic needle lung biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Haseem Ashraf, Lørenskog, Select A State, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zaetta JM, Licht MO, Fisher JS, Avelar RL; Bio-Seal Study Group. A lung biopsy tract plug for reduction of postbiopsy pneumothorax and other complications: results of a prospective, multicenter, randomized, controlled clinical study. J Vasc Interv Radiol. 2010 Aug;21(8):1235-43.e1-3. doi: 10.1016/j.jvir.2010.04.021. PMID 20656223
- [Background] Ahrar JU, Gupta S, Ensor JE, Mahvash A, Sabir SH, Steele JR, McRae SE, Avritscher R, Huang SY, Odisio BC, Murthy R, Ahrar K, Wallace MJ, Tam AL. Efficacy of a Self-expanding Tract Sealant Device in the Reduction of Pneumothorax and Chest Tube Placement Rates After Percutaneous Lung Biopsy: A Matched Controlled Study Using Propensity Score Analysis. Cardiovasc Intervent Radiol. 2017 Feb;40(2):270-276. doi: 10.1007/s00270-016-1489-9. Epub 2016 Nov 8. PMID 27826786
- [Background] Grage RA, Naveed MA, Keogh S, Wang D. Efficacy of a Dehydrated Hydrogel Plug to Reduce Complications Associated With Computed Tomography-guided Percutaneous Transthoracic Needle Biopsy. J Thorac Imaging. 2017 Jan;32(1):57-62. doi: 10.1097/RTI.0000000000000247. PMID 27870824